CLINICAL TRIAL: NCT00597233
Title: Comparative Evaluation of Human NPH Insulin + Insulin Aspart and Human NPH Insulin + Human Soluble Insulin in Type 1 Diabetes Mellitus
Brief Title: Human Insulin NPH and Insulin Aspart in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1529
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin aspart
Drug: soluble human insulin
Drug: insulin NPH

SUMMARY:
This trial is conducted in South America. This aim of this trial is to evaluate the comparative prandial blood glucose lowering profile in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Treatment with insulin NPH
* Body Mass Index (BMI) below 30 kg/m2

Exclusion Criteria:

* Total daily insulin dose greater than 1.40 IU/kg
* Treatment with oral antidiabetic drugs (OADs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2002-10; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Prandial blood glucose lowering profile | between 1st and 2nd post prandial hours

SECONDARY OUTCOMES:
Hypoglycaemic events
Adverse events
Serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Junín, Argentina

REFERENCES:
- [Result] Cintora H, Rodrigues M, Klyver MI, Claus-Hermerg H, González G, Kanevsky D, Medrano G, Sánchez A. Insulina Aspártica versus insulina soluble humana: Estudio comparativo cruzado en pacientes con diabetes tipo 1. Revista de la Sociedad Argentina de Diabetes 2004; 38 (4): 218-224
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com